CLINICAL TRIAL: NCT07221344
Title: A Phase 1/2a Placebo-Controlled Dose-Escalating Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ARO-MAPT-SC in Healthy Subjects and Subjects With Early Alzheimer's Disease
Brief Title: Study of ARO-MAPT-SC in Healthy Subjects and Subjects With Early Alzheimer's Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AROMAPT-SC-1001
Record Dates: First submitted 2025-10-23; First posted 2025-10-27 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease; Alzheimer Disease, Early Onset
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ARO-MAPT-SC (Experimental): ARO-MAPT-SC injection
  Interventions: Drug: ARO-MAPT-SC
- Placebo (Placebo Comparator): Sterile normal saline (0.9%)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ARO-MAPT-SC — • single or multiple doses of ARO-MAPT-SC by subcutaneous (SC) injection
  Arms: ARO-MAPT-SC
Drug: Placebo — • calculated volume to match active treatment by SC administration
  Arms: Placebo

SUMMARY:
Study to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics of ARO-MAPT-SC compared to placebo in adult healthy volunteers and in participants with early Alzheimer's disease (AD), defined as mild cognitive impairment due to AD and mild AD dementia.

ELIGIBILITY:
Inclusion Criteria (All Participants):

* Body mass index between 18.0 and 35.0 kg/m^2 at Screening
* Not pregnant or breast-feeding
* Able and willing to provide written informed consent prior to the performance of any study specific procedures
* Participants of childbearing potential must agree to use highly effective contraception in addition to a condom during the study and for at least 90 days following the end of the study or last dose of study drug, whichever is later; participants must not donate sperm or eggs during the study and for at least 90 days following the end of the study or last dose of study drug whichever is later

Inclusion Criteria (Alzheimer's Disease):

* Adults aged 50 to 75 years of age with a clinical diagnosis of early AD and plasma, CSF, or imaging biomarkers consistent with the diagnosis
* On stable doses of AD-related medications for at least 8 weeks prior to Screening Visit and throughout the Screening period until Day 1

Exclusion Criteria (All Participants):

* Uncontrolled hypertension
* Human immunodeficiency virus (HIV) infection (seropositive at Screening)
* Seropositive for hepatitis B (HBV) or hepatitis C (HCV) at Screening
* Intellectual disability or significant behavioral neuropsychiatric manifestation
* Clinically significant cardiac, liver, or renal disease
* Any contraindications to lumbar puncture

Note: Additional inclusion/exclusion criteria may apply per protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) Over Time | Through End of Study (EOS), Day 270

SECONDARY OUTCOMES:
PK of ARO-MAPT-SC: Maximum Observed Plasma Concentration (Cmax) | Through 48 hours postdose
PK of ARO-MAPT-SC: Time to Maximum Plasma Concentration (Tmax) | Through 48 hours postdose
PK of ARO-MAPT-SC: Area Under the Plasma Concentration (AUC) Versus Time Curve From Time Zero to 24 Hours (AUC0-24) | Through 24 hours postdose
PK of ARO-MAPT-SC: AUC Versus Time Curve From Time Zero to 48 Hours (AUC0-48) | Through 48 hours postdose
PK of ARO-MAPT-SC: AUC Versus Time Curve From Time Zero to the Last Quantifiable Plasma Concentration (AUC0-t) | Through 48 hours postdose
PK of ARO-MAPT-SC: AUC Versus Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) | Through 48 hours post-dose
PK of ARO-MAPT-SC: Apparent Terminal Elimination Half-life (t1/2) | Through 48 hours postdose
PK of ARO-MAPT-SC: Apparent Systemic Clearance (CL/F) | Through 48 hours postdose
PK of ARO-MAPT-SC: Apparent Terminal-phase Volume of Distribution (Vz/F) | Through 48 hours postdose
PK of ARO-MAPT-SC: Amount Excreted (Ae) of Unchanged Drug in Urine From Time Zero to 24 Hours Postdose | Through 24 hours postdose
PK of ARO-MAPT-SC: Percentage of Administered Drug Recovered (Fe) in Urine From Time Zero to 24 Hours Postdose | Through 24 hours postdose
PK of ARO-MAPT-SC: Renal Clearance (CLR) | Through 24 hours postdose
Change from Baseline in Total Protein in Cerebral Spinal Fluid (CSF) Over Time | Baseline through EOS, Day 270
Change from Baseline in Glucose in CSF Over Time | Baseline through EOS, Day 270
Change from Baseline in Cell Count in CSF Over Time | Baseline through EOS, Day 270

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site 1, Grafton, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No